CLINICAL TRIAL: NCT02932826
Title: Phase 1/ Phase 2 Study of the Therapeutic Effect of Ex-vivo Expanded Umbilical Cord Blood Regulatory T Cells on Autoimmune Diabetes
Brief Title: Safety Study and Therapeutic Effects of Umbilical Cord Blood Treg on Autoimmune Diabetes
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Zhiguang Zhou, MD/PhD, Second Xiangya Hospital of Central South University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015CX009
Record Dates: First submitted 2016-10-11; First posted 2016-10-13 (Estimated); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Autoimmune Diabetes; Umbilical Cord Blood Cell; Regulatory T Lymphocyte; Cell Therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treg Treatment + Insulin (Experimental): subjects will be treated with Umbilical Cord Blood Regulatory T cells Therapy and insulin according to routine clinical practice at the discretion of the treating physician
  Interventions: Biological: Umbilical Cord Blood Regulatory T cells Therapy; Drug: Insulin
- Insulin (Active Comparator): subjects will be treated with insulin according to routine clinical practice at the discretion of the treating physician
  Interventions: Drug: Insulin

INTERVENTIONS:
Biological: Umbilical Cord Blood Regulatory T cells Therapy — Receive Treg infusion: 1~5*10^6/kg b.w. in 100ml NS
  Arms: Treg Treatment + Insulin
Drug: Insulin — Treated according to routine clinical practice at the discretion of the treating physician

SUMMARY:
The purpose of this study is to investigate the safety and therapeutic effect of ex-vivo expanded umbilical cord blood regulatory T cells on autoimmune diabetes.

DETAILED DESCRIPTION:
The regulatory T cells (Treg) used in this study will be produced from human umbilical cord blood. The umbilical cord blood will be freshly collected and immediately separated to buffy coat in a GMP laboratory, thus to be further sorted into Treg and other subsets. Then the Treg will be expanded ex-vivo for approximately 14 days until tested for its surface markers and suppressive ability. During the time of ex-vivo expansion, eligible autoimmune diabetes patients will be recruited and admitted to our hospital in order to go through required examinations. Once the Treg product has reached the safety and efficacy standards, the patient will receive the Treg product infusion under close surveillance of doctors and then go through regular follow-ups to investigate the safety and therapeutic effect of the Treg product on autoimmune diabetes patients.

ELIGIBILITY:
Inclusion Criteria:

1. Autoimmune diabetes patients are screened for enrollment in the study if both clinical signs and laboratory tests meet the diagnosis standards of American Diabetes Association
2. Diagnosis of Autoimmune Diabetes within 3 years of screening
3. Between 6 to 60 years of age
4. Positive for at least one of the anti-islet autoantibodies: GADA, IA2A, ZnT8A
5. Fasting or postprandial plasma C-peptide more than 200 pmol/L
6. Written informed consent from the patient or the patient's parents for patients under the age of 18 years

Exclusion Criteria:

1. Any clinically significant diseases in liver (ALT and AST over 2 times upper normal limit), kidney (Scr over 133umol/L), and heart
2. Presence of anemia (Hb ≤100g/L), leukopenia (<3.5×10^9/L)
3. Presence of disorder in coagulation or anticoagulation, or thrombocytopenia (platelets <100×10^9/L)
4. Presence of acute metabolic disorders; In the case of acute ketone acidosis, with blood ketone over 0.3mmol/L and pH lower than 7.30
5. Presence of any kind of chronic infection or immune deficiency, including hepatitis B, hepatitis C, HIV, syphilis or tuberculosis
6. Chronic use of systemic glucocorticoids or other immunosuppressive agents for over 3 months
7. Any history of malignancy
8. Female patients who are pregnant or breastfeeding; any female who is unwilling to use a reliable and effective form of contraception for 2 years afer recruitment
9. Presence of any infectious diseases, including active skin infections, flu, fever, upper or lower respiratory track infections; those who wish to participate in the study should keep the infection under control for at least 1 week before receiving Treg product infusion
10. Presence of diabetic microvascular or macrovascular diseases
11. Presence of hypertension
12. Any medical condition that, in the opinion of the investigator, will interfere with safe participation in the trial

Ages: 6 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-10; Primary Completion 2025-06 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse events as a Measure of Safety and Tolerability | 2 years
  The number of participants with adverse events, laboratory abnormalities and other signs of toxicity. Particular focus will be on the number and severity of infusion reactions, complications related to infection, and any potential negative impact on the course of diabetes.

SECONDARY OUTCOMES:
C-peptide | 2 years
  Measure the C-peptide level of participant after treatment
Insulin requirement | 2 years
  Measure the Insulin requirement of participant after treatment
Blood glucose | 2 years
  Measure the blood glucose level of participant after treatment
HbA1c | 2 years
  Measure the HbA1C level of participant after treatment
Autoimmune Status | 2 years
  The autoimmune status refers to the state and degree of autoimmune attacks in autoimmune diabetes patients. Measures include change in titer of autoantibodies, change in subsets of immune cells, and change in autoimmune related cytokines.

CONTACTS AND LOCATIONS:
Overall Officials: Zhiguang Zhou, MD/PhD, Principal Investigator — Second Xiangya Hospital of Central South University
Locations (1):
- Institute of Metabolism and Endocrinology, Second Xiangya Hospital, Central South University, Changsha, Hunan, China

REFERENCES:
- [Background] Milward K, Issa F, Hester J, Figueroa-Tentori D, Madrigal A, Wood KJ. Multiple unit pooled umbilical cord blood is a viable source of therapeutic regulatory T cells. Transplantation. 2013 Jan 15;95(1):85-93. doi: 10.1097/TP.0b013e31827722ed. PMID 23263503
- [Background] Fan H, Yang J, Hao J, Ren Y, Chen L, Li G, Xie R, Yang Y, Gao F, Liu M. Comparative study of regulatory T cells expanded ex vivo from cord blood and adult peripheral blood. Immunology. 2012 Jun;136(2):218-30. doi: 10.1111/j.1365-2567.2012.03573.x. PMID 22348606
- [Background] Brunstein CG, Miller JS, Cao Q, McKenna DH, Hippen KL, Curtsinger J, Defor T, Levine BL, June CH, Rubinstein P, McGlave PB, Blazar BR, Wagner JE. Infusion of ex vivo expanded T regulatory cells in adults transplanted with umbilical cord blood: safety profile and detection kinetics. Blood. 2011 Jan 20;117(3):1061-70. doi: 10.1182/blood-2010-07-293795. Epub 2010 Oct 15. PMID 20952687